CLINICAL TRIAL: NCT00809107
Title: Cryopreserved-Thawed Embryo Transfer in Natural Cycle or in Natural Cycles Controlled by External Administration of hCG: a Prospective Randomized Study
Brief Title: Frozen Embryo Transfer (FET) in Natural Cycles or in Natural Cycles Controlled by Human Chorionic Gonadotropin (hCG) Administration
Acronym: FRET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Kyrou Dimitra, centre of reproductive medicine-UZ
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC3471
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Infertility
Keywords: natural cycle; FET; spontaneous LH pic; HCG
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HCG GROUP
  Interventions: Drug: HCG
- 2 (No Intervention): LH pick

INTERVENTIONS:
Drug: HCG — 5000IU
  Other Names: pregnyl
  Arms: 1

SUMMARY:
The rational of the study is to assess the implantation, pregnancy and live birth rates after the transfer of frozen- thawed embryos in natural cycles with spontaneous Luteinizing Hormone (LH)/Progesterone rise or in natural cycles controlled by human chorionic gonadotropin (hCG) for final oocyte maturation and ovulation.

ELIGIBILITY:
Inclusion Criteria:

* age <40
* BMI:18-29Kg/m2
* day 3 embryo transfers
* previously IVF or ICSI

Exclusion Criteria:

* irregular cycles
* oocyte donation cycles

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-07 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Implantation rate | 2 years

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Reproductive Medicine, Brussels, Belgium

REFERENCES:
- [Background] Gelbaya TA, Nardo LG, Hunter HR, Fitzgerald CT, Horne G, Pease EE, Brison DR, Lieberman BA. Cryopreserved-thawed embryo transfer in natural or down-regulated hormonally controlled cycles: a retrospective study. Fertil Steril. 2006 Mar;85(3):603-9. doi: 10.1016/j.fertnstert.2005.09.015. PMID 16500326